CLINICAL TRIAL: NCT02021435
Title: Using Salt Substitute to Reduce Population Blood Pressure in Tibet: Tibet Salt Reduction Study
Brief Title: Tibet Salt Reduction Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: The George Institute for Global Health at PUHSC (Unknown); The George Institute for Global Health, Australia (Other); Science and Technology Department of Ningxia (Unknown); People's Hospital of Tibet (Unknown); People's Hospital of Maizhokunggar (Unknown); Tibet University (Other); Peking University (Other); People's Hospital of Damxung County, Tibet (Unknown)
Responsible Party: Principal Investigator, Xingshan Zhao, Vice-president; Director, Department of Cardiology, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013BAI05B04
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Blood Pressure; Cardiovascular Diseases; Death
MeSH Terms: conditions — Cardiovascular Diseases; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salt Substitute (Experimental): salt substitute
  Interventions: Dietary Supplement: salt substitute
- Control (No Intervention): Participants continue to buy salt at their own expense

INTERVENTIONS:
Dietary Supplement: salt substitute — Free salt substitute provided
  Arms: Salt Substitute

SUMMARY:
1. Research background

   - High blood pressure is one of the most important risk factors to cardiovascular diseases (CVDs). Reducing population blood pressure can control CVD incidence and lower mortality effectively. Much research has proven that adjusting for Na and K intake level can reduce blood pressure. According to the China Salt Substitute Study, the systolic blood pressure of intervention group which used salt substitute is 5.4 mmHg lower than that of control group. Life expectancy in Tibet is 67 years old. It is estimated that the use of salt substitute among population in Tibet can reduce total mortality in Tibet by 20%. China Salt Substitute Study in Tibet (CSSS-Tibet), found that salt substitute is effective in lowering both systolic and diastolic blood pressure and offers a simple, low-cost approach for hypertension control among Tibetans in China (unpublished results). However, the study focused on hypertensive patients, the effectiveness of hypertension control by providing free salt substitute to the entire population remains unknown, and a large-scale trial is needed.
2. Objectives

   - Primary objective is to observe the effect of providing salt substitute on population blood pressure in Tibet. Secondary objective is to observe the effect of such intervention on population mortality, cardiovascular mortality and life expectancy. In addition, the data collected from high-risk population (sub-group) in the study will be used in China Salt Substitute and Stroke Study (SSaSS). Also, serum cholesterol and random blood glucose of people over 60 in Tibet will be collected.
3. Method

   * The study is a open, cluster-randomized, controlled trial.
   * 30 villages with 15 to 35 households each and a distance of at least five kilometers in between will be selected from Damxung county and Maizhokunggar county. The two counties have an average altitude of over 4000 meters in Tibet Autonomous Region.
   * All selected villages will be randomly assigned to intervention group or control group on a 1:1 ratio.
   * All household in the selected villages will be recruited if they meet the eligibility criteria. Approximately 4,500 participants will be enrolled
   * Intervention group receives free salt substitute. Control group will continue to buy their own normal salt. Both group will receive the same health education on salt reduction.
4. Outcome - Primary outcome is blood pressure. Secondary outcomes include total mortality, cardiovascular disease mortality, life expectancy, serum cholesterol level of people over 60, and random blood glucose level of people over 60.

ELIGIBILITY:
Inclusion Criteria:

* All family households in the selected satellite village will be invited to participate in the study

Family households will be excluded from participating if they meet one or more of the following exclusion criteria:

* Any member in the family is using a potassium-sparing diuretic
* Any member in the family is using a potassium supplement
* Any member in the family has serious renal impairment
* Any member in the family over 18 could not sign informed consent
* Life expectancy of any member in the family is shorter than 6 months in doctor's opinion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline in blood pressure between intervention and control | Baseline, 6,12, 24 months

SECONDARY OUTCOMES:
Difference in total mortality between intervention and control | 6, 12, 24 months
Difference in cardiovascular disease mortality between intervention and control | 6,12, 24 months
Difference in life expectancy between intervention and control group | 6, 12, 24 months
The distribution of blood glucose level in population over 60 years old | baseline
Distribution of serum cholesterol level in population over 60 years old | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xingshan Zhao, M.D., Principal Investigator — Beijing Jishuitan Hospital
Locations (2):
- China (2):
  - Damxung, Tibet
  - Maizhokunggar, Tibet